CLINICAL TRIAL: NCT01066897
Title: Imaging the Nucleus Accumbens in Major Depressed Patients 'Treated With Pramipexole
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of funding prevented further recruitment
Sponsor: Stanford University (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Principal Investigator, Jennifer Keller, Principle Investigator, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SU-02042010-4902; 17847
Record Dates: First submitted 2010-02-09; First posted 2010-02-10 (Estimated); Results first posted 2017-05-16 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-04

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Pramipexole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pramipexole (Experimental): Patients will receive 0.125 mg of pramipexole three times a day for the first week, 0.25 mg three times a day for the second week, and 0.5 mg three times a day for the third week. The dose will then be adjusted as needed by the treating physician (Dr. DeBattista), with a target range of 1.0 mg to 1.5 mg per day. Dose escalations will continue until 1) achievement of the primary endpoint (> 50% reduction from baseline on the HDRS scores; 2) intolerable side effects; or 3) completion of the 8-week study. Participants will be seen weekly the first four weeks and biweekly thereafter. Side effects, depression, and anhedonia will assessed at each visit.
  Interventions: Drug: Pramipexole
- Healthy Controls (No Intervention): Non depressed, non-intervention comparison group

INTERVENTIONS:
Drug: Pramipexole — Patients will received increasing dose of pramipexole
  Arms: Pramipexole

SUMMARY:
We hope to learn how a brain circuit that is important to the understanding of depression, anhedonia and positive affect responds to a novel pharmaceutical treatment for depression and related symptoms. Adults who have a diagnosis of major depression and are not completely responsive to antidepressant medication will be sought out for participation; as will an equal number of adults not suffering from the disorder. Those suffering from depression will be given pramipexole, an investigational medication for eight weeks during which information will be collected about mood, cognition, and brain function. Adults not suffering from depression will also be evaluated with these measures.

DETAILED DESCRIPTION:
Patients who meet DSM-IV criteria for major depression(using the SCID),have a Hamilton Depression Rating Scale score of at least 18, and who are not complete responders to antidepressant medications will be invited to participate in an open label study with pramipexole. Patients who are not complete responders to an adequate trial of an antidepressant (see inclusion criteria below) will be openly treated with pramipexole for 8 weeks. Participants must be between the ages of 20-55 and will include both men and women. Patient's mood will be assessed each visit using the Hamilton Depression (HDRS) and will also complete a series of questionnaires. This will include the physical and social anhedonia scales (Chapman et al., 1976; Eckblad et al., 1982), the Snaith-Hamilton Pleasure Scale (SHAPS; Franken et al., 2007; Snaith et al., 1995), the Mood and Anxiety Symptom Questionnaire Short Form (MASQ; Watson, Weber, et al., 1995; Watson, Clark, et al., 1995), and the Positive and Negative Affect Scale (Watson & Clark, 1991)among others. No other adjunctive agents will be allowed during the eight weeks of the study. Patients will be seen for four weeks on a weekly basis, then biweekly thereafter.

Patients will receive 0.125 mg of pramipexole three times a day for the first week, 0.25 mg three times a day for the second week, and 0.5 mg three times a day for the third week. The dose will then be adjusted as needed by the treating physician (Dr. DeBattista), with a target range of 1.0 mg to 1.5 mg per day. Dose escalations will continue until 1) achievement of the primary endpoint (> 50% reduction from baseline on the HDRS scores; 2) intolerable side effects; or 3) completion of the 8-week study. Participants will be seen weekly the first four weeks and biweekly thereafter. Side effects, depression, and anhedonia will assessed at each visit.

Depressed participants will also undergo functional MRI and neuropsychological testing twice, once at baseline and once after completion of the medication. 20 healthy control subjects with no history of Axis I disorders and who score less than 5 on the HDRS will participate in the baseline MRI, neuropsychological testing, and clinical ratings/questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Must meet DSM-IV criteria for Major Depressive Disorder
2. HAM-D score >18 on a 21-item assessment at eligibility
3. On at least an adequate dose of fluoxetine (40 mg/day), paroxetine (40 mg/day) paroxetine CR (50mg), sertraline (150 mg/day), citalopram (40 mg/day), escitalopram (20 mg/day), venlafaxine (150 mg/day), mirtazapine (30 mg/day), or duloxetine (60 mg/day) for at least 6 weeks (monotherapy).
4. 20-55 years of age

Exclusion Criteria:

1. Substance abuse in the past 6 months
2. ECT in the past 6 months
3. On a MAOI, tricyclic antidepressant, lithium, an antipsychotic, thyroid augmentation, 2 antidepressants simultaneously or lamotrigine
4. History of any psychosis including psychotic depression
5. History of Bipolar I, Bipolar II, or Bipolar NOS illness, or concurrent symptoms of mania or hypomania that do not meet the criteria for any bipolar disorder
6. History of compulsive gambling
7. Pregnant females or females of childbearing years not using adequate birth control in the opinion of the investigators
8. Known sensitivity to Pramipexole
9. Significant suicide risk in the opinion of the investigators
10. Significant medical conditions that would preclude safe participation in the study in the opinion of the investigators
11. Psychoactive drugs other than one of the antidepressants listed on Inclusion criteria #4. (A non-barbiturate sedative or hypnotic or benzodiazepine such as trazodone 50mg/day, zolpidem 10mg/day, lorazepam 3mg/day or clonazepam 2mg/day will be allowed if it has been in use for at least 1 month prior to the baseline visit.)
12. Significant abnormalities are observed in screening laboratory evaluation.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Keller, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Controls: Non depressed, non treatment comparison group
Period: Overall Study
Arm/Group | Pramipexole | Healthy Controls
Started | 7 | 9
Completed | 5 | 9
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — stopped study after developing the flu. | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Healthy Controls: Non depressed, non treatment comparison group from baseline
- Total: Total of all reporting groups
Arm/Group | Pramipexole | Healthy Controls | Total
Number analyzed (Participants) | 7 | 9 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.00 (14.12) | 34.78 (14.0) | 38.81 (14.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 10
  Male | 0 | 6 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 7 | 5 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 9 | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Discontinued Study Due to Side-effects of the Medication
Time Frame: throughout the 8 weeks
Population: # of participants who dropped out due to medication side-effects
Measure: Count of Participants; unit: Participants
Arm/Group | Pramipexole | Healthy Controls Who Did Not Take Medication
Number analyzed (Participants) | 7 | 9
Participants | 2 | 0
Statistical Analysis 1: Comparison: Pramipexole vs Healthy Controls Who Did Not Take Medication; Test type: Other; p = .002, Chi-squared

2. Primary Outcome: % Change in Hamilton Depression Rating Scale From Baseline to week8
Description: Utilized the Hamilton Depression Rating Scale, 21-item version to assess depressive symptoms, with a range of 0-63. Higher scores equals more depression. For the change score, where higher equals greater improvement in depressive symptoms.
  Healthy controls were not utilized in this analysis, as no week 8 ratings for health controls were obtained.
Time Frame: Baseline and weeks 8
Population: For two drop outs, used LOCF
Measure: Mean (Standard Deviation); unit: percentage reduction in depression score
Arm/Group | Pramipexole
Number analyzed (Participants) | 7
percentage reduction in depression score | .46 (.42)
Statistical Analysis 1: Comparison: Pramipexole; For the 2 dropouts, used LOCF; Test type: Superiority or Other; p = .067, t-test, 2 sided; One sample t-test to determine if the % change in HAMD was different from 0; Mean Difference (Net) = .368, Standard Deviation .44

3. Primary Outcome: Change in Mesolimbic Reward System Activity From Pre to Post Treatment (8 Weeks)
Description: Because of the limited number of depressed patients who completed the study (n=5) and noisy/unusable imaging data at various time points, this data was unable to be examined.
Time Frame: baseline and Week 8
Population: Because of the limited number of depressed patients who completed the study (n=5) and noisy/unusable imaging data at various time points, this data was unable to be examined.
Arm/Group | Pramipexole | Healthy Controls
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Mesolimibic Reward Activity Baseline Differences in Depression vs Healthy Controls
Description: Because of the small number of depressed patients and noisy/unusable data, analyses were not run.
Time Frame: Baseline
Population: Because of the small number of depressed patients and noisy/unusable data, analyses were not run.
Arm/Group | Pramipexole | Healthy Controls
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From date of randomization, every two weeks, assessed up to 8 weeks. Adverse events were only collected for the pramipexole group.
Arm/Group | Pramipexole
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 2/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pramipexole (N=7)
somnolence (Nervous system disorders) | 1 (2)
nausea (Nervous system disorders) | 1 (1)
restless leg (Nervous system disorders) | 1 (1)
odd thoughts (Psychiatric disorders) | 1 (1)
insomnia (Nervous system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The sample size is really too small for statistical analyses. Lack of funding prevented further recruitment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No